CLINICAL TRIAL: NCT02642003
Title: To Assess the Efficacy of Granulocyte Colony Stimulating Factor Versus Standard Medical Therapy in Patients of Decompensated Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ashish Kumar, Co investigator, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gastro-2014-OL
Record Dates: First submitted 2015-12-21; First posted 2015-12-30 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-04

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Granulocyte Colony-Stimulating Factor

ARMS (2):
- GCSF+SMT (Experimental): 5-day course of GCSF (5 μg/kg/d) plus standard medical therapy for 6 months
  Interventions: Drug: Granulocyte Colony Stimulating Factor
- SMT (No Intervention)

INTERVENTIONS:
Drug: Granulocyte Colony Stimulating Factor
  Arms: GCSF+SMT

SUMMARY:
Background and Aims: Liver transplantation is the only curative treatment modality for decompensated cirrhosis and is limited by donor organ availability and financial resources; thus many patients die while awaiting liver transplant. Granulocyte colony stimulating factor (GCSF) therapy can mobilize bone marrow stem cells for tissue regeneration, and has been shown to benefit patients with liver disease. The investigators evaluated the efficacy of GCSF therapy in decompensated cirrhosis in an open labelled randomized control trial.

Patients and Methods: Consecutive patients with decompensated cirrhosis of mixed etiologies were randomized to receive either a 5-day course of GCSF (5 μg/kg/d) plus standard medical therapy for 6 months (Group-A); or standard medical therapy alone for 6 months (Group-B). At the end of 6 months their survival were compared.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to75 years
* Patients of decompensated cirrhosis with CTP ≥6 and ≤ 13
* Liver transplantation not feasible soon (due to financial reasons or unavailability of donors).

Exclusion Criteria:

* Hepatocellular Carcinoma
* Sepsis (Any culture positive: blood, urine, any other obvious source of infection: UTI, SBP): Patients were included after sepsis is controlled.
* Any organ failure
* Grade 3 or 4 Hepatic Encephalopathy, Active Variceal bleed, Hepatorenal Syndrome: Patients might be included after clinical improvement
* HIV seropositivity
* Pregnancy
* Refusal to participate in the study
* Previous known hypersensitivity to G-CSF

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of participants alive at 6 months | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology & Hepatology, Sir Ganga Ram Hospital, New Delhi, New Delhi, India

REFERENCES:
- [Derived] Prajapati R, Arora A, Sharma P, Bansal N, Singla V, Kumar A. Granulocyte colony-stimulating factor improves survival of patients with decompensated cirrhosis: a randomized-controlled trial. Eur J Gastroenterol Hepatol. 2017 Apr;29(4):448-455. doi: 10.1097/MEG.0000000000000801. PMID 27930386